CLINICAL TRIAL: NCT05537597
Title: Repetitive Transcranial Magnetic Stimulation for Musculoskeletal Pain in Patients With Parkinson's Disease：Efficacy and Safety, Electrophysiological Mechanisms and Influence on Motor and Other Non-motor Symptoms
Brief Title: Repetitive Transcranial Magnetic Stimulation for Musculoskeletal Pain in Patients With Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Cheng-Jie Mao, Associate Professor, Second Affiliated Hospital of Soochow University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JD-LK-2021-132-01
Record Dates: First submitted 2022-09-02; First posted 2022-09-13 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Parkinson's Disease; Musculoskeletal Pain; Repetitive Transcranial Magnetic Stimulation; Primary Motor Cortex; Electroencephalography; Neuromodulation
MeSH Terms: conditions — Parkinson Disease; Musculoskeletal Pain

STUDY DESIGN:
Intervention Model Description: Patients will be randomised to receive either active or sham-rTMS according to a 2:1 ratio.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The figure-of-eight coils used for active or sham stimulation are similar, including the emitted sound and the scalp tapping sensation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M1-rTMS group (Experimental)
  Interventions: Procedure: active M1-rTMS
- sham-rTMS group (Sham Comparator)
  Interventions: Procedure: sham rTMS

INTERVENTIONS:
Procedure: active M1-rTMS — Magnetic stimulation will be carried out using a MagPro X100 machine with a MCF-B70 figure-of-eight coil (Magventure, Farum). All rTMS sessions will be assisted by a neuronavigation system (TMS Navigator，Localite GmbH), maintaining the M1 target and the orientation of coil stable during stimulation sessions. The M1 target was defined as the "hand knob" region, which corresponds to the motor cortical representation of the hand, regardless of the location of pain.
  Stimulation paradigm consists of 20 trains of pulses with an intra-train frequency of 20 Hz, resulting in 2000 pulses for a total duration of 20 minutes.
  The stimulation intensity will be 80% of RMT, defined as the lowest stimulation intensity necessary to induce a visible muscle twitch of the hand contralateral to the stimulated hemisphere.
  Participants will receive 7 sessions of treatment once a day in the same time continuously for 7 days, and keep antiparkinsonism drugs unchanged throughout the whole study.
  Arms: M1-rTMS group
Procedure: sham rTMS — The sham protocol was similar to the rTMS protocol. Sham stimulations will be performed with a MCF-P-B65 figure-of-eight coil (Magventure) to M1, assisted by a neuronavigation system.
  The following stimulation parameters will be used: stimulus frequency 20 Hz; stimulus intensity 80 % of RMT; total stimulation pulses 2,000; total stimulation time 20 min.
  Participants will receive 7 sessions of treatment once a day in the same time continuously for 7 days, and keep antiparkinsonism drugs unchanged throughout the whole study.
  Arms: sham-rTMS group

SUMMARY:
Pain is an increasingly recognized non-motor symptom of Parkinson's disease (PD), with significant prevalence and negative impact on the quality of life of patients.

Repetitive transcranial magnetic stimulation (rTMS) of the primary motor cortex（M1）has been proposed to provide definite analgesic effect for pain syndromes. However, very few placebo-controlled studies have been performed specifically to relieve pain in PD. What's more, based on behavioral measures alone, it is impossible to reveal the full network dynamics reflecting the impact of TMS.

Electroencephalography (EEG), with high temporal resolution, records signal that its origin in electrical neural activity, which makes it suitable for measuring TMS-evoked activation. By recording the TMS induced neuronal activation directly from the cortex, TMS-EEG provides information on the excitability, effective connectivity of cortical area, thus exploring cortical network properties in different functional brain states. In addition, the use of EEG offers great prospects as a tool to select the right patients in order to achieve adequate, long-term pain relief.

Besides assessing the efficacy and safety of high-frequency neuronavigated M1-rTMS in PD patients with musculoskeletal pain, the objective of this study additionally aimed to characterize cortical activation behind pain relief. Influence on motor and other non-motor symptoms after rTMS were also investigated.

DETAILED DESCRIPTION:
Pain can appear as a pre-motor symptom, and its intensity could be severe enough to be the dominant non-motor symptom in the course of PD patients.

It estimated the prevalence of painful phenomena in PD to be 30 to 85% (mean 66%), which is significantly greater than the age-matched general population. Painful experiences in PD are highly heterogeneous and complex, which is difficult to describe for patients but also diagnose for neurologists. In addition, this common and disabling symptom receives inadequate analgesic treatment.

The distinction between these pain subtypes is required so that different therapeutic strategies can be established for each type of pain. The King's Parkinson's Pain scale (KPPS) was validated to identify and rate the various types of pain in PD. Fourteen items cover seven main domains, including musculoskeletal pain, chronic body pain (central or visceral), fluctuation-related pain, dyskinetic-dystonic pain, nocturnal pain, oro-facial pain, discolouration/oedema/swelling, and radicular pain. Of these subtypes, musculoskeletal pain is common.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation technique that may be useful for the treatment of various psychiatric and neurological disorders. The mechanisms underlying rTMS effects remain to be elucidated.

rTMS is postulated to induce neuronal excitability changes in a set of cortical and subcortical areas involved in pain processing and modulation. Interestingly, M1 stimulation had a positive effect on brain structures that are related to the affective-emotional components of pain, such as the insular cortex and cingulate cortex.

The best efficacy for chronic pain has been achieved when primary motor cortex (M1) is stimulated at high frequency (5 to 20 Hz, 80% of the resting motor threshold (RMT)), as in previous rTMS studies in analgesia.

In TMS, time-varying magnetic fields generates electrical currents in the cortex. TMS pulses can either directly or trans-synaptically depolarize neurons, and these neural activities can be recorded through the skull by EEG electrodes placed on the scalp. The combination of TMS with simultaneous EEG can be used to assess excitability, inhibition, plasticity and connectivity across almost all areas of the cortical mantle.

The characterization of potential TMS-EEG predictors and markers could be the theoretical basis for verifying the response to neuromodulation protocols.

In this randomised, double-blind, placebo-controlled study, the efficacy and safety of 7 sessions of 20 Hz-rTMS delivered to M1 will be assessed in PD patients with chronic musculoskeletal pain.

A single-pulse TMS-EEG and resting-state EEG directly provide information on the cortical mechanisms before and after rTMS of M1.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic PD was diagnosed according to the 2015 Movement Disorder Society (MDS) clinical diagnostic criteria
2. Hoehn and Yahr stages of I to III
3. musculoskeletal pain was detected based on the Ford classification system for pain in PD，chronic pain for ≥3 months
4. stable antiparkinsonian therapy for ≥4 weeks

Exclusion Criteria:

1. Contraindications to rTMS
2. unstable ongoing psychiatric disorder, history of substance abuse (alcohol, drugs)
3. histories of deep brain stimulation surgery
4. Mini-mental State Examination scores ≤24
5. Other pain conditions, such as apparent osteoarthritis, or rheumatoid arthritis depended on laboratory or imaging findings

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline over 2 months (group by time interaction) in KPPS | before the first rTMS session (day 1), after rTMS therapy at day8、1month、2month
  King's PD Pain Scale (KPPS) includes 14 items rating the severity and frequency of pain, each item scored by severity (0-3) multiplied by frequency (0-4), resulting in a subscore of 0 to 12, with a total possible score range from 0 to 168.
Change from baseline over 2 months (group by time interaction) in MKPPS | before the first rTMS session (day 1), after rTMS therapy at day8、1month、2month
  Modified King's PD Pain Scale (MKPPS)，the modified version which is more suitable for Chinese people, combined with Ford's pain subtypes basing on the original. It covers five main domains, including 16 items, each item scored by severity (0-3) multiplied by frequency (0-4), resulting in a total possible score range from 0 to 192.
Change in pain intensity scores (VAS) | before the first rTMS session (day 1), after rTMS therapy at day8、1month、2month
  VAS, a 0-10 numeric rating scale with 0= no pain and 10=maximal pain
Adverse event | through study completion, an average of 2 month
  Any adverse events occurred and the reasons leading to treatment discontinuation will be recorded. The severity and relevance will be rated as mild, moderate or serious by investigators.

SECONDARY OUTCOMES:
Changes in resting-state EEG oscillations | before the first rTMS session (day 1), after rTMS therapy (day8)
  During EEG recordings, participants will sit alone in a quiet room and be requested to minimize any other body movements, mostly with eyes closed.
  We will use a TMS-compatible EEG amplifier (neuracle, changzhou, China) and a cap (Greentek, Wuhan, China) providing 64 TMS-compatible coated-electrodes with positions of the international 10/20 system.
  The signals recorded will be digitized at a sampling rate of 1kHz. Skin/electrode impedance will be maintained below 10KΩ. The EEG recording protocol consists of a 5-min resting-state paradigm without any task involvement.
Changes in Resting-State EEG Functional Connectivity | before the first rTMS session (day 1), after rTMS therapy (day8)
  The functional connectivity of the identified brain region showing significant difference of cortical oscillations will be further investigated.
Alterations of TMS-elicited evoked potentialspotentials | before the first rTMS session (day 1), after rTMS therapy (day8)
  Single-pulse TMS of the M1 will be performed during EEG recording by means of a figure-of-eight coil oriented to elicit posterolateral-anteromedial current flow in the brain. The signal was sampled at 16 kHz. Participants will wear inserted earplugs to avoid signals contamination by the click associated with the TMS discharge.
  the interval of each sTMS will be set at 4 seconds to avoid habituation with repeated stimulation.
  Each participant will undergo a 20-min session about 120 TMS trials at intensity of 120%RMT.
Changes in PD-Motor Symptoms Scale total score | before the first rTMS session (day 1), after rTMS therapy at day8、1month、2month
  The participants will be evaluated in their "ON" medication states. The scales used to assess motor symptoms are parts III (ranging from 0 to 132) and IV (ranging from 0 to 24) of the MDS-Unified PD Rating Scale (MDS-UPDRS), with higher scores indicating more severe symptoms.
Changes in PD-Non-Motor Symptoms Scale total score | before the first rTMS session (day 1), after rTMS therapy at day8、1month、2month
  The participants will be evaluated in their "ON" medication states. The scales used to assess non-motor symptoms included parts I (ranging from 0 to 52) and II (ranging from 0 to 52) of the MDS-UPDRS, with higher scores indicating more severe symptoms.
Changes in PD depression score | before the first rTMS session (day 1), after rTMS therapy at day8、1month、2month
  The depression score (ranging from 0 to 76 with higher scores indicating more severe depression) from the 24 items Hamilton Depression Scale (HAMD).
Changes in PD anxiety score | before the first rTMS session (day 1), after rTMS therapy at day8、1month、2month
  The anxiety score (ranging from 0 to 60 with higher scores indicating more severe anxiety) from the 14 items Hamilton Anxiety Scale (HAMA).
Changes in PD autonomic Symptoms score | before the first rTMS session (day 1), after rTMS therapy at day8、1month、2month
  The Scale for Outcomes in Parkinson's disease for Autonomic Symptoms (SCOUP-AUT, maximal score 67, with higher scores indicating higher autonomic nervous system dysfunction).
Changes in PD sleep problem score | before the first rTMS session (day 1), after rTMS therapy at day8、1month、2month
  The sleep problem index (from 0 to 68 with higher scores indicating more severe sleep problem) from the PD Sleep Scale-2 (PDSS-2).
Changes in PD daytime sleepiness score | before the first rTMS session (day 1), after rTMS therapy at day8、1month、2month
  The daytime sleepiness will be assessed by the Epworth Sleeping Scale (ESS), maximal score 24, with higher scores indicating more severe symptoms.
Changes in PD quality of life score | before the first rTMS session (day 1), after rTMS therapy at day8、1month、2month
  We will also assess change in quality of life from the Parkinson's Disease Questionnaire-39 (PDQ-39), ranging from 0 to 156 with higher scores indicating more serious influence.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valkovic P, Minar M, Singliarova H, Harsany J, Hanakova M, Martinkova J, Benetin J. Pain in Parkinson's Disease: A Cross-Sectional Study of Its Prevalence, Types, and Relationship to Depression and Quality of Life. PLoS One. 2015 Aug 26;10(8):e0136541. doi: 10.1371/journal.pone.0136541. eCollection 2015. PMID 26309254
- [Background] Silverdale MA, Kobylecki C, Kass-Iliyya L, Martinez-Martin P, Lawton M, Cotterill S, Chaudhuri KR, Morris H, Baig F, Williams N, Hubbard L, Hu MT, Grosset DG; UK Parkinson's Pain Study Collaboration. A detailed clinical study of pain in 1957 participants with early/moderate Parkinson's disease. Parkinsonism Relat Disord. 2018 Nov;56:27-32. doi: 10.1016/j.parkreldis.2018.06.001. Epub 2018 Jun 6. PMID 29903584
- [Background] Chaudhuri KR, Rizos A, Trenkwalder C, Rascol O, Pal S, Martino D, Carroll C, Paviour D, Falup-Pecurariu C, Kessel B, Silverdale M, Todorova A, Sauerbier A, Odin P, Antonini A, Martinez-Martin P; EUROPAR and the IPMDS Non Motor PD Study Group. King's Parkinson's disease pain scale, the first scale for pain in PD: An international validation. Mov Disord. 2015 Oct;30(12):1623-31. doi: 10.1002/mds.26270. Epub 2015 Jun 11. PMID 26096067
- [Background] Picarelli H, Teixeira MJ, de Andrade DC, Myczkowski ML, Luvisotto TB, Yeng LT, Fonoff ET, Pridmore S, Marcolin MA. Repetitive transcranial magnetic stimulation is efficacious as an add-on to pharmacological therapy in complex regional pain syndrome (CRPS) type I. J Pain. 2010 Nov;11(11):1203-10. doi: 10.1016/j.jpain.2010.02.006. Epub 2010 Apr 28. PMID 20430702
- [Background] O'Connell NE, Marston L, Spencer S, DeSouza LH, Wand BM. Non-invasive brain stimulation techniques for chronic pain. Cochrane Database Syst Rev. 2018 Apr 13;4(4):CD008208. doi: 10.1002/14651858.CD008208.pub5. PMID 29652088
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449